CLINICAL TRIAL: NCT06986265
Title: Association of Cachexia and Gut Microbiome in Dialysis Patients : Investigation of the Interactions With Uremic Toxins and Inflammation.
Brief Title: CKD Cachexia and Gut Microbiome
Acronym: DYNAMICA
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); FRC- Fonds de la Recherche Clinique (Unknown); SFNDT - Société Francophone de Néphrologie, Dialyse et Transplantation (Unknown)
Responsible Party: Sponsor
Other Study IDs: B403202400099
Record Dates: First submitted 2024-12-05; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Diseases; Cachexia
Keywords: cachexia; Protein energy wasting; microbiota; chronic kidney disease; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dialysis patients: Collection of clinical data and biological samples
  Interventions: Other: Collection of clinical data and biological sampling

INTERVENTIONS:
Other: Collection of clinical data and biological sampling — Multiple measures relevant to cachexia, such as body weight, body mass index (BMI), muscle mass (handgrip strength using a Jamar hand dynamometer, mid-upper arm muscle circumference), appetite (Functional Assessment of Anorexia/Cachexia Therapy [FAACT], Simplified Nutritional Appetite Questionnaire [SNAQ], Automated Self- Administered Dietary Assessment Tool [ASA24]) will be recorded at inclusion (T0), after 6 months (T6) and after one year of follow-up (T12). Body composition will be assessed by bioelectrical impedance analysis at T0, T6 and T12, and by CT-scan at T0 and T12. In parallel, gut microbiota composition on feces collection will be determined at the two time points (T0 and T12). Markers of systemic and intestinal inflammation will be assessed at T0 and T12. Serum levels of uremic toxins will be measured at T0 and T12. Human muscle biopsies will be performed at the time of a surgical intervention.

SUMMARY:
Cachexia is common in patients with chronic kidney disease (CKD) and is associated with increased morbidity and mortality. Cachexia is a complex syndrome, in which inflammation and retention of uremic toxins are two main contributing factors. In this context, the role of the gut microbiome in CKD cachexia and the potential benefit of increasing the dialysis dose have been poorly explored. Here the investigators propose to study the links between cachexia and the gut microbiome, in association with inflammation and uremic toxins, in dialysis.

The specific objectives are the followings:

1. Set up a prospective cohort of deeply characterized kidney failure patients treated with hemodialysis (in-center, self-care dialysis in a satellite unit and at home) and peritoneal dialysis, including evaluation of cachexia, body composition, collection of feces and blood to characterize the gut microbiota, measure serum levels of uremic toxins and inflammatory markers, with a longitudinal follow-up.
2. To compare cachectic versus non-cachectic dialysis patients in terms of gut microbiota, inflammatory markers, level of uremic toxins, muscle transcriptome, dialysis dose and modality. In a subgroup analysis, the investigators plan to compare the different techniques of dialysis (in-center vs home-hemodialysis vs peritoneal dialysis).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of kidney failure (stage V)
* Maintenance dialysis for at least 3 months
* Understanding of the trial procedures and ability to adhere to the trial protocol

Exclusion Criteria:

* Severe nonadherence to the dialysis procedure
* Life expectancy below 1 year
* Chronic inflammatory disease of the digestive tract (Crohn's disease, ulcerative colitis)
* Bariatric surgery
* Active cancer
* Pregnancy
* Antibiotics consumption in the month preceding the inclusion
* Gastro-intestinal surgery, colonoscopy, or probiotics consumption in the 3 months preceding the inclusion
* Drugs influencing body composition initiated ≤ 1 month : systemic corticosteroids, anabolic drugs as insulin or testosterone, post-menopausal hormone therapy, injectable contraceptives.
* Known endocrinological disorders potentially leading to hypo- or hypermetabolism, untreated or treated for ≤ 1 month : disorders of thyroid gland, adrenal glands...
* Patients under weight loss drugs : GLP1 agonists, orlistat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population studied is adult kidney failure patients treated with hemodialysis (in-center, self-care dialysis in a satellite unit or at home) or with peritoneal dialysis for more than 3 months.
  The principal investigator, who is a Nephrologist and works at the Nephrology Department, in Cliniques universitaires Saint-Luc, in contact with dialysis patients, will check patient eligibility, collect the consent from the subjects who agree to participate and allocate an ID number.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Composition and function of the gut microbiota | Throughout the entire study, approximately during 5 years
  Sequencing DNA extracts from patients' feces to obtain the description of gut microbiota composition and function

SECONDARY OUTCOMES:
Level of inflammatory markers | Throughout the entire study, approximately during 5 years
Level of uremic toxins | Throughout the entire study, approximately during 5 years
Metabolomics profile | Throughout the entire study, approximately during 5 years
Dialysis dose | Throughout the entire study, approximately during 5 years
  number of hours of dialysis per week
Dialysis modality | Throughout the entire study, approximately during 5 years
  in-center hemodialysis vs self-care dialysis in a satellite unit vs home-hemodialysis vs peritoneal dialysis
Body composition | Throughout the entire study, approximately during 5 years
  Bioelectrical impedance analysis (in kg)
Body composition | Throughout the entire study, approximately during 5 years
  Noncontrast enhanced CT scan of the abdomen at the level of the third lumbar vertebra (L3)
Quality of life | Throughout the entire study, approximately during 5 years
  FAACT (Functional Assessment of Anorexia-Cachexia Therapy) and FACIT (Functional Assessment of Chronic Illness Therapy - Fatigue Scale) questionnaires
Handgrip strength | Throughout the entire study, approximately during 5 years
  Jamar dynamometer (in kg)
Physical activity | Throughout the entire study, approximately during 5 years
  International Physical Activity Questionnaire (IPAQ)
Appetite | Throughout the entire study, approximately during 5 years
  Simplified Nutritional Assessment Questionnaire (SNAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Inès Dufour, MD, Principal Investigator — Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels
  - UCLouvain, Brussels

IPD SHARING:
Plan to Share IPD: No